CLINICAL TRIAL: NCT03775018
Title: Transversus Abdominis Plane (TAP) Blockade as Multimodal Analgesia for Pain Control in One-Anastomosis Gastric Bypass (OAGB)
Brief Title: TAP Blockade for Pain Control in One-Anastomosis Gastric Bypass
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Department of Surgery, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HRJC 18-14
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The analgesic treatment applied will be blinded to the treatment and to the epidemiology nurse who will assess the postoperative pain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversus abdominis plain blockade (Experimental): The patients will undergo Transversus abdominis plain blockade, associated with intravenous analgesia
  Interventions: Procedure: Transversus abdominis plane blockade; Drug: Intravenous analgesia
- Intravenous analgesia (Active Comparator): The patients will receive intravenous analgesia with Acetaminophen (1g/6h)
  Interventions: Drug: Intravenous analgesia

INTERVENTIONS:
Procedure: Transversus abdominis plane blockade — Patients will undergo Transversus abdominis plane blockade with Bupivacaine 0.25% 30ml, applied in the plane between the internal oblique muscle and the trasnversus abdominis. The injection will be performed laterally to the port-sites, bilaterally at the same levels.
  Arms: Transversus abdominis plain blockade
Drug: Intravenous analgesia — Acetaminophen 1g/6h iv will be administered

SUMMARY:
Patients will be randomized into 2 groups:

* TAP: Patients undergoing TAP blockade, associated with intravenous Acetaminophen analgesia
* IV: Patients receiving only intravenous Acetaminophen analgesia

Postoperative pain 24 hours after surgery will be evaluated.

DETAILED DESCRIPTION:
Patients will be randomized into 2 groups:

* TAP: Patients undergoing TAP blockade, associated with intravenous Acetaminophen analgesia (1g/6h)
* IV: Patients receiving only intravenous Acetaminophen analgesia (1g/6h)

Postoperative pain 24 hours after surgery will be evaluated, by a Visual Analogic Scale (VAS), ranging from 0 to 100mm.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing One-anastomosis gastric bypass (OAGB) as primary bariatric procedure

Exclusion Criteria:

* Patients undergoing OAGB as revisional procedure
* Patients undergoing other bariatric procedures
* Patients undergoing additional surgical procedures during the same surgical act (band removal, cholecystectomy, hernioplasty, or hiatal hernia treatment)
* Patients with history of allegy to local anesthetic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2018-12-13 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Pain will be assessed 24 hours after surgery by a Visual Analogic Scale, ranging from 0 to 100mm

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia, MD, PhD, Study Director — Hospital Rey Juan Carlos